CLINICAL TRIAL: NCT02968316
Title: Bioelectric Impedance Analysis and Pregnancy Outcomes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maternal Fetal Medicine Associates (Other)
Responsible Party: Principal Investigator, Nathan Fox, Physician, Maternal Fetal Medicine Associates
Other Study IDs: 1
Record Dates: First submitted 2016-11-14; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: all consecutive pregnant women presenting for prenatal care
  Interventions: Other: BIA measurement

INTERVENTIONS:
Other: BIA measurement — observation only

SUMMARY:
This is a prospective observational study correlating Body Impedance Analysis (BIA) with pregnancy outcomes.

DETAILED DESCRIPTION:
BIA is a new method of measuring total body water, fat, and lean mass. It is measured noninvasively, and the investigators plan on using the InBody analyzer (www.InBody.com) in this study. The analysis takes a few seconds and only requires the participant to stand on a small platform and grasp a small device in each hand. The machine then uses low electrical current to analyze the body composition and produce a read-out.

The investigators plan on doing this analysis longitudinally across gestation in multiple trimesters to analyze the ability to predict maternal morbid conditions prior to the current clinically-based criteria as a novel marker to aid in routine prenatal care, as compared to the traditional weight measurement currently being done.

Both increased maternal prepregnancy weight (body mass index) and increased maternal gestational weight gain have been associated with increased risks of multiple obstetrical complications (both maternal and fetal). The investigators seek to compare the current standard with BIA in its ability to predict maternal/fetal adverse outcomes such as gestational diabetes, preeclampsia, and cesarean delivery.

PRIOR RESEARCH

There are a few studies in pregnant patients correlating BIA and pregnancy outcomes:

1. Sween et al performed BIA on 370 women and found that body fat composition correlated with the development of preeclampsia.
2. Gomes de Silva et al performed BIA in 65 women with preeclampsia and 51 controls and found that BIA results differed between the two groups.
3. Marshall et al performed BIA on 41 pregnant women in the third trimester as part of a multimodal analysis of body composition
4. Xu et al correlated BIA with the onset of gestational diabetes

PROTOCOL

* Patients in this MFM practice will be approached at the time of their initial pregnancy visit and asked to participate.
* If they agree and sign informed consent, the following will occur:

  * The participant's name will be placed on a list of participants
  * The participant will have an InBody analysis performed by one of the office nurses or medical assistants. The results will not be shared with the participant nor the treating physicians. Rather, the results will be filed until after the participant delivers.
  * Participants will have the InBody analysis performed in each trimester at the time of scheduled office visits as well as at the post-partum visit, which is routinely scheduled at approximately 6 weeks after delivery. Those results will also not be shared with the participants or physicians.
  * After the postpartum visit, the data from the InBody analysis will be entered into a de-identified database, along with the participant's baseline characteristics, pregnancy events, and delivery outcomes, all of which are already in the participant's office chart. No personal identifiers will be required for the database. The data will be used to correlate InBody results with pregnancy outcomes.
  * The only identifier will be the actual list of participants, which is required to plan for who needs InBody analysis during their prenatal visit.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women

Exclusion Criteria:

* refusal to participate

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Preeclampsia | from date of enrollment up to 6 weeks after delivery (within 1 year)
gestational diabetes | from date of enrollment up to 6 weeks after delivery (within 1 year)
cesarean delivery | from date of enrollment up to delivery (within 1 year)
neonatal birth weight | from date of enrollment up to delivery (within 1 year)
gestational age at delivery | from date of enrollment up to delivery (within 1 year)

CONTACTS AND LOCATIONS:
Locations (1):
- Maternal Fetal Medicine Associates, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No